CLINICAL TRIAL: NCT06379009
Title: Evaluating the Effect of a Structured Home-based Physical Training Program for Kidney Transplant Recipients With Impaired Pre-transplant Physical Function
Brief Title: Effect of Home-based Training Program for Kidney Transplant Recipients (HOMETRAIN-KTR)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: South-Eastern Norway Regional Health Authority (Other)
Responsible Party: Principal Investigator, Tommy Aronsen, Nephrologist/phd-student, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 473076
Record Dates: First submitted 2024-04-15; First posted 2024-04-23 (Actual); Last update posted 2024-04-24 (Actual); Status verified 2024-04

CONDITIONS: Kidney Transplant; Complications; Frailty; Physical Disability
Keywords: Training
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Intervention Model Description: 2 arms randomized control study. The intervention arm is exposed of a 12 week home-based training program. The control arm follow standard of care.
Masking Description: Both participants and investigators will know which arm the participants are randomized to. Training is not easy to mask
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Home-based training (Experimental): Structured home-based training program over 12 week period (in addition to standard care). The program has been prepared by physiotherapists and starts 4 weeks after kidney transplantation. It consists of 2 sessions of strength training and 1 session of cardio training each week. In addition, optional training sessions on the other days of the week. The patients will be followed up by phone every week, heart rate monitor and patients logs. A physiotherapist will guide the patients in the beginning of the intervention period
  Interventions: Other: Training
- Standard of care (No Intervention): This group will undergo standard physical training program in addition to standard care. They will be informed about the importance of regular exercise after discharge from hospital.

INTERVENTIONS:
Other: Training — 12 week home-based training program
  Arms: Home-based training

SUMMARY:
Does home-based training work in kidney transplant recipients with reduced physical function?

The goal of this clinical trial is to learn if home-based training works to better physical function in adult kidney transplant recipients. It will also learn about participants preoperative physical function. The main question it aim to answer is

* Does home-based training improves physical function in kidney transplant recipients.
* All the participants are assessed to have reduced physical function before the transplantation

Participants will:

* follow either a home-based training program or todays standard of physical activity after kidney transplantation
* the program starts 4 weeks after the transplantation and lasts for 12 weeks. A physiotherapist will help the participants in the beginning.
* the program consists of both cardio-training, strength-straining and optional activity
* the training group will be followed up every week by phone. Their activity will be documented via patients logs and heart rate monitor.
* the effect of the training will be evaluated one year after the transplantation

DETAILED DESCRIPTION:
Title:

Evaluating the effect of a structured home-based physical training program for kidney transplant recipients with impaired pre-transplant physical function (HOMETRAIN KTR)

Background and Aims:

Frailty and impaired physical function are prevalent among patients undergoing kidney transplantation (KTx), and is an independent risk factor for poor outcome after transplantation. Limited number of studies have prospectively investigated the efficacy of exercise training for KTx-recipients with low pre-transplant physical function. Our aim is to evaluate the effect of a structured 12 week home-based physical training program delivered to recipients with low pre transplant physical function, on physical function and frailty at 1-year post transplant.

Method:

HOMETRAIN-KTR is a 2-arm unblinded Norwegian clinical trial with RCT design. Patients will be recruited at admission for KTx at Oslo University Hospital, Rikshospitalet. Patients who score below 60 at 36-Item Short Form Survey will be included and tested with 6-minute walking test, Clinical Frailty Scale, hand-grip strength, 30 seconds Sit-to-Stand test, and questionnaire about physical activity and psychological distress. Included patients are randomized to either training group or control group (standard of care). The training group will, under supervision by a physiotherapist, start a 12-week structured home-based training program from week 4 post-KTx. The training program consist of a combination of strength training, cardio training and optional activities. During the intervention period, the intervention group will receive regular follow-up by phone. The training sessions will be documented via patients logs and heart rate monitor. At one year post-KTx, all patients will undergo the same tests as at inclusion.

Inclusion of patients will start in January 2024, and continue for the next 2-3 years. The investigators aim to include 200 patients, 100 in each arm. The study will evaluate physical function, frailty, graft function, patient survival, HRQoL and physiological distress during the time-span of the study.

Hypothesis:

The HOMETRAIN-KTR study is supposed to bring new knowledge about the effect of a physical training program on frail KTx-recipients. Such information is highly relevant to improve KTx outcomes and to optimize the utilization of the limited source of donor organs.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years old or older and going through Ktx
* Scores 75 or lower at physical function at SF-36 at time of KTx
* Able to perform the 6MWT
* Able to speak, read and understand Norwegian or English
* Being mentally and cognitively capable of participating in the intervention and responding to follow-up questionnaires

Exclusion Criteria:

- none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-01-01 (Estimated)

PRIMARY OUTCOMES:
6-minute walking distance test | Baseline and after 52 weeks
  Test of physical function. How many meters the patient manage to walk in 6 minutes.
Clinical Frailty Scale | Baseline and after 52 weeks
  Test for frailty. Validated test for this purpose. Score 1-9. The higher the score the more frail

SECONDARY OUTCOMES:
Hand-grip strength | Baseline, week 7, week 26 and week 52
  Using a hand-dynamometer to measure hand-grip strength. Average of 3 trials
30 seconds Sit-to-stand test | Baseline, week 7, week 26 and week 52
  Get up from chair. Number of repetitions in 30 seconds
Bone density test | Week 7 and week 52
  Dual-energy X-ray absorptiometry (DXA)
Bioelectrical impedance phase angle to measure muscle mass and strength. | Week 7 and 52
  Measuring bioelectrical impedance phase angle with a machine called BWA 2,0 Body. Water Analyzer. Phase angle is an indicator of muscular death, and is inversely related to muscle mass and strength in frail subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Marit Helen Andersen, Principal Investigator — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No